Efficacy of Kinesio Taping in Musculoskeletal Neck Pain in Short and Medium Term. A Randomized Control Double Blinded Clinical Trial. Guillermo Ceniza-Bordallo et al. 1 June 2021. University Complutense of Madrid.





## Efficacy of Kinesio Taping in Musculoskeletal Neck Pain in Short and Medium Term. A Randomized Control Double Blinded Clinical Trial

<u>TITLE:</u> Efficacy of Kinesio Taping in Musculoskeletal Neck Pain in Short and Medium Term. A Randomized Control Double Blinded Clinical Trial

INVESTIGATOR PRINCIPAL: GUILLERMO CENIZA-BORDALLO

**PROJECT ENTITIES:** COMPLUTENSE UNIVERSITY OF MADRID & NURSERY, PHYSIOTHERAPY AND PODIATRY FACULTY.

## **NUMBER OF IDENTIFIACTION:**

**DATE:** 1<sup>ST</sup> JUNE 2021.

Efficacy of Kinesio Taping in Musculoskeletal Neck Pain in Short and Medium Term. A Randomized Control Double Blinded Clinical Trial. Guillermo Ceniza-Bordallo et al. 1 June 2021. University Complutense of Madrid.





## **Statistical Analysis Plan**

The statistical software IBM SPSS® (Statistical Package for the Social Sciences 22, SPSS Inc., Chicago, IL USA) was used. The quantitative variables were presented as mean ± standard deviation (SD), while the qualitative variables were shown as an absolute value (relative frequency percentage). To study the effects produced on the main variables of each intervention at different times of evaluation, an analysis of variance of repeated measures (factorial ANOVA) was applied. Secondarily, the same analysis was performed for each intervention on the secondary variable.

Additionally, the effect size (partial eta squared,  $\eta 2$ ) was calculated for the changes produced by comparing within the same intervention group (intragroup) and comparing between intervention groups (intergroup), following the classification criteria described by Cohen: small (0.1 - 0.24), moderate (0.25 - 0.39), and large (> 0.4)

The interpretation of the statistical tests was performed based on a significance level of 5% (p <0.05) for a 95% confidence interval.